CLINICAL TRIAL: NCT05974943
Title: The Effect of Problem Solving And Decision Making Education On Problem Solving and Decision Making Skills of Nurse Managers
Brief Title: The Effect of Problem Solving and Decision Making Training Given to Nurses Managers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Berra YILMAZ KUŞAKLI, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 92450
Record Dates: First submitted 2023-06-09; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Nurse; Problem Solving; Decision Making; Education
Keywords: nurse manager; problem solving; decision making; education

STUDY DESIGN:
Intervention Model Description: These studies aimed to enable the evaluation of nurse managers' problem-solving and decision-making abilities from the perspective of their subordinates. The study was carried out using a systematic and randomized controlled design, incorporating elements such as pre-test-post-test, experimental, and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the pre-post training and 3rd-month evaluations of problem-solving skills of the nurse managers in (Experimental): The research was conducted with randomized control, pretest-posttest, experimental, and control group design. By using G*Power analysis, it was determined that the experimental group of the nurse managers was 30 people and included randomly in the sample calculation of the study. The experimental group was given 2 days of problem-solving and decision-making training. Before the training, the nurse administrators in the experimental group were administered the Participant Information Form-Nurse Manager, PSI, DMSS and two Case Evaluation Forms and Problem Solving and Decision Making Information Form-Pre-Test-Post-Test.
  Interventions: Other: Problem Solving And Decision Making Education
- the pre-post training and 3rd-month evaluations of the decision-making skills of the nurse managers (No Intervention): The research was carried out in randomized control, pretest-posttest, experimental and control group design. In the sample calculation of the study, 30 of the manager nurses were determined by using G*Power analysis as the control group and were included randomly. No intervention was made in the control group. At the same time as the experimental group, the nurse administrators in the control group were also administered the Participant Information Form-Nurse Manager, PSI and DMSS.
- pre-training and 3rd-month evaluations of regarding the problem-solving and decision-making skills (No Intervention): Three months after the initial assessment, the nurse managers in the experimental and control groups were administered PCI and CVSQ.

INTERVENTIONS:
Other: Problem Solving And Decision Making Education — The Problem-Solving and Decision-Making Training Program, which was based on developing problem-solving and decision-making skills of nurse managers in the experimental group (n=30), was prepared. 2 faculty members and the researcher organized the training program consisting of four modules and 16 hours.
  In the content of the Training Program; the definition of the concept of problem-solving and decision-making, the process of problem-solving and decision-making and decision-making models, the impact of decision-making on employee, patient and organizational outcomes, and the importance of managers' roles in decision-making, the importance of the role of nurse managers in decision making, the impact of managerial decisions on patient care outcomes, the impact of managerial decisions on nurse outcomes, the impact of administrative decisions on organizational results/performance, problem-solving, and decision-making techniques and case studies.
  Arms: the pre-post training and 3rd-month evaluations of problem-solving skills of the nurse managers in

SUMMARY:
This research was conducted to evaluate the impact of the Problem Solving and Decision Making Training program, which was developed to enhance the problem-solving and decision-making skills of nurse managers at the lower, middle, and upper levels, by the subordinates and superiors of nurse managers. To assess the problem-solving and decision-making skills of nurse managers as perceived by their subordinates, the Problem-Solving Inventory-Managerial Version (PSI-MV) and Decision-Making Styles Scale-Managerial Version (DMSS-MV) underwent adaptation, validity, and reliability studies. These studies aimed to enable the evaluation of nurse managers' problem-solving and decision-making abilities from the perspective of their subordinates.

DETAILED DESCRIPTION:
This research was conducted to evaluate the impact of the Problem Solving and Decision Making Training program, which was developed to enhance the problem-solving and decision-making skills of nurse managers at the lower, middle, and upper levels, by the subordinates and superiors of nurse managers. To assess the problem-solving and decision-making skills of nurse managers as perceived by their subordinates, the Problem-Solving Inventory-Managerial Version (PSI-MV) and Decision-Making Styles Scale-Managerial Version (DMSS-MV) underwent adaptation, validity, and reliability studies. These studies aimed to enable the evaluation of nurse managers' problem-solving and decision-making abilities from the perspective of their subordinates. The study was carried out using a systematic and randomized controlled design, incorporating elements such as pre-test-post-test, experimental, and control groups. In the initial phase of the research, the target population comprised 2,108 nurses employed at a city hospital in Istanbul, while the actual sample included 328 nurses. The validity and reliability studies of PSI-MV and DMSS-MV were carried out. In the scale analyses, psycholinguistic and psychometric properties were examined. In the second part of the research, a sample of 300 nurses, including 60 nurse managers and their subordinates (30 in the experimental group and 30 in the control group), was included using G*Power analysis for sample calculation.

ELIGIBILITY:
Inclusion Criteria:

The criteria for inclusion in the sample for nurse managers were determined as follows:

* Working as a nurse manager,
* Working in a managerial position for at least six months,
* Volunteering to participate in the research,
* Ensuring full-time participation in the training program to be held within the scope of the research for the experimental group.

Inclusion criteria for subordinate nurses or nurse managers were determined as follows:

* Working under a nurse manager in the experimental or control group,
* Working with the nurse manager he/she evaluated for at least six months,
* Volunteer to participate in the research.

Exclusion Criteria:

* Not meeting the sampling inclusion criteria,
* Filling the data collection tools incompletely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
The change in the Decision-Making Styles Scale | up to 1 week
The decrease in the mean score of the Problem Solving Inventory | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Betül SÖNMEZ, Ass.pr.dhd, Principal Investigator — drhembetulsonmez@gmail.com
Locations (1):
- İstanbul Üniversitesi - Cerrahpaşa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2024 and unlimited
Access Criteria: This work, which is a doctoral thesis, can be accessed after it is published at https://tez.yok.gov.tr/UlusalTezMerkezi/.
URL: https://tez.yok.gov.tr